CLINICAL TRIAL: NCT04104724
Title: A Feasibility Study of a Compassion-focused Self-help Intervention Designed to Increase Access to Cervical Screening Following Sexual Assault
Brief Title: CFT Self-Help for Accessing Cervical Screening After Sexual Assault
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Holloway University (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Jane Smallwood, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSmallwoodDClinPsy
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Trauma, Psychological; Sexual Violence; Cervical Cancer
MeSH Terms: conditions — Psychological Trauma; Uterine Cervical Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help (Experimental): Immediate access to self-help materials
  Interventions: Other: Self-help
- Control (No Intervention): Wait-list control - treatment as usual (no intervention)

INTERVENTIONS:
Other: Self-help — self-help materials - cognitive behavioural and compassion-focused; psychoeducation, practical help re. attending cervical cancer screening
  Other Names: compassion-focused therapy; cognitive behaviour therapy; psychoeducation
  Arms: Self-help

SUMMARY:
The aim of this study is to evaluate the feasibility of a new self-help intervention designed to support individuals (anyone with a cervix) to access cervical cancer screening following the experience of sexual assault, by addressing psychological barriers identified by previous research, specifically shame, low self-efficacy and the re-traumatising nature of attending to sexual health after sexual trauma.

DETAILED DESCRIPTION:
The study aims to investigate the acceptability, feasibility and limited efficacy of a discrete, easily accessed (mobile phone, tablet or computer) self-help intervention to support people to access cervical screening independently.

The study will use a wait-list control design, with participants randomly allocated to receive access to the intervention immediately or after a six-week wait.

The intervention will be in the form of a web app and will contain a range of psychoeducational material and practice exercises following a cognitive-behavioural and compassion-focused approach to understanding and coping with trauma, building self-compassion and increasing confidence in ability to attend and complete a screening.

ELIGIBILITY:
Inclusion Criteria:

* Has a cevix
* Within age range for cervical cancer screening in UK (25-64 years)
* Experience of sexual assault (in childhood and/or adulthood; not within last 12 months)
* Currently experiencing difficulty attending cervical cancer screening
* Has access to smartphone/computer with internet
* Has a valid email address
* Able to read and understand English
* Living in UK

Exclusion Criteria:

* No cervix
* Outside of UK cervical cancer screening age range
* No experience of sexual assault or sexual assault occurred within last 12 months
* No access to smartphone or computer and internet
* Unable to read or understand English
* Not living in UK
* In acute mental health crisis

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2020-05-03 (Estimated); Study Completion 2020-05-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability: Is the intervention acceptable to the intended audience? | Six weeks
  A series of statements written by the researchers asking for feedback on the intervention, including frequency of use, interest in the content, satisfaction. To be rated on a five-point scale (Completely agree - Completely disagree). This will be analysed descriptively (e.g. how many people would recommend the app to others having similar difficulties?)
Behavioural change - Does use of the intervention lead to an increase in bookings and attendance at screenings? | Six weeks
  Participants will be asked to report their progress at baseline and follow-up by answering a series of questions written by the researchers, for example 'I have contacted my GP surgery to ask them when cervical screening clinics take place' - Yes/No; 'I attended my cervical screening appointment' - Yes/No.
Behavioural change - Does use of the intervention facilitate completing a cervical screening? (i.e. does the intervention have limited efficacy?) | Six weeks
  Participants will be asked whether or not they have completed their cervical screening at baseline and follow-up. Answer options will be yes/no/appointment booked but hasn't happened yet

SECONDARY OUTCOMES:
Psychological change - Does use of the intervention lead to increased self-efficacy and self-compassion, and reduced shame? | Six weeks
  Experience of Shame Scale - Items scored from 1-4 (not at all - very much); higher scores indicate higher levels of shame. Total score ranges from 25-100; can also be broken down into subscales: characterological (range 12-48), behavioural (range 9-36) and bodily (range 4-16) shame.
  The Compassionate Engagement and Action Scale - Self-Compassion subscales. All items scored on a scale of 1-10 (Never-Always), total scores range from 10-100 with a higher score indicating greater self-compassion.
  Self-efficacy scale - questions to assess self-efficacy specifically relating to ability to attend a cervical screening (e.g. 'I can contact my GP surgery to book a cervical screening') - to be rated on a scale of 0 (cannot do at all) to 100 (highly certain can do), leading to an overall total ranging from 0 to 1200; higher scores suggest greater self-efficacy.
Psychological change - distress | Six weeks
  Additional clinical outcome measures will be the PCL-5, measuring PTSD symptomatology; the PHQ-2, measuring low mood and the GAD-2, measuring anxiety. On each of these measures higher scores suggest more distress.
  Items on the PCL-5 are scored from 0 (not at all) to 4 (extremely) with a possible total range from 0 to 80. The PHQ-2 and GAD-2 each comprise two items scored from 0 (not at all) to 3 (nearly every day) with possible total scores ranging from 0 to 6.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews B, Qian M, Valentine JD. Predicting depressive symptoms with a new measure of shame: The Experience of Shame Scale. Br J Clin Psychol. 2002 Mar;41(Pt 1):29-42. doi: 10.1348/014466502163778. PMID 11931676
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Gilbert, P., Catarino, F., Duarte, C., Matos, M., Kolts, R., Stubbs, J., ... & Basran, J. (2017). The development of compassionate engagement and action scales for self and others. Journal of Compassionate Health Care, 4(1), 4.
- [Background] Bandura, A. (2006). Guide for constructing self-efficacy scales. Self-efficacy Beliefs of Adolescents, 5(1), 307-337.
- [Background] Cadman L, Waller J, Ashdown-Barr L, Szarewski A. Barriers to cervical screening in women who have experienced sexual abuse: an exploratory study. J Fam Plann Reprod Health Care. 2012 Oct;38(4):214-20. doi: 10.1136/jfprhc-2012-100378. PMID 23027982
- See also: My Body Back Project — http://mybodybackproject.com